CLINICAL TRIAL: NCT01145586
Title: A Phase III, Non-Inferiority, Randomized, Blind, Parallel-Group, Multicentre, Multiple-Dose, Comparative Clinical Study of Lactase Eurofarma and Lactaid®, Assessing the Efficacy and Safety in the Treatment of Patients With Lactose Intolerance"
Brief Title: A Non-inferiority, Multicenter and Randomized, Multiple-Dose Study About a Treatment to Hypolactasia
Acronym: LAILAII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF099-2
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — Lactase

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactase EUF (Experimental): 1 oral tablet of the test drug before breakfast, lunch and dinner for 42 consecutive days
  Interventions: Drug: Lactase Oral Tablets
- Lactase Ref (Active Comparator): 1 oral tablet of the comparative drug before breakfast, lunch and dinner for 42 consecutive days
  Interventions: Drug: Lactase Oral Tablets

INTERVENTIONS:
Drug: Lactase Oral Tablets — 3 tablets/day for 42 days Take with breakfast, lunch and dinner

SUMMARY:
The primary objective is to determine the compared clinical efficacy of Lactase Eurofarma (test drug), showing non-inferiority to Lactaid® (comparative drug) in the supportive treatment of lactose intolerance and to assess the safety and tolerance of Lactase Eurofarma (test drug) in the supportive treatment of lactose intolerance.

ELIGIBILITY:
Inclusion Criteria:

* To have participated in the single-dose clinical study (EF099) previously performed, with the clinical response being considered as satisfactory by the investigator
* The patient should be a male or female, aged between 18 and 60 years old
* Have a medical history consistent with lactose intolerance, confirmed by the test of hydrogen in the expired air
* The female patients should agree to use birth control methods during the study participation
* To be able to meet the study instructions and all the visits required
* To give a free consent to participate in the study and sign the informed consent form (ICF).

Exclusion Criteria:

* Smoking
* Secondary hypolactasia
* Gastrointestinal inflammatories diseases - present diverticular disease, diabetic gastropathy or neoplasias
* Colonoscopy or colon cleaning procedure 4 weeks before the start of study
* Latrogenic: unnoticed intake of laxatives in over-the-counter drugs or alternative medicine, intake of cereal bran or probiotics
* Diagnosis of HIV, immunodepression of any origin, or cancer under treatment.
* Diagnosis of other comorbidity that, at the investigator's discretion, may compromise the study participation (e.g., systemic infection during the study or use of antibiotics in the last 4 weeks, diabetes mellitus, uncontrolled hypertension or renal failure),
* Hypersensitivity or previous laboratory or clinical adverse event related to the use of lactase or any of the components of the formulations used in the study
* Incapacity to understand and complete the study questionnaires, including the questions that require the use of the Visual Analogue Scale and ICF
* Pregnancy or lactation
* Use of alcohol, exceeding 3 doses daily
* Participation in another clinical study on the last 12 months
* Patient having some chronic pulmonary disease that, in the investigator's opinion, may harm or interfere with the expired hydrogen test (e.g., cystic fibrosis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Hydrogen value in the expired air | 03 times
  Hydrogen value in the expired air for 3h after the patient exposure to the standardized Lactose 25g dose with interventional exogenous Lactase (comparative and test drugs).

SECONDARY OUTCOMES:
Signs and Symptoms Diary | 42 days
  * Signs and Symptoms Diary, registered for the period between V0 and V1 / V1 and V2;
  * The Specific Symptom Score registered during the tests of hydrogen in the expired air;
  * Global Evaluation of the Treatment Tolerance by the patient and the investigator; Frequency of adverse events noted.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Machado, M.D, Principal Investigator — Hospital São Lucas / PUCRS; Heda Amarante, M.D, Principal Investigator — Hospital Nossa Senhora das Graças; Sender Miszputen, M.D, Principal Investigator — Hospital São Paulo/UNIFESP; Wilson Catapani, M.D, Principal Investigator — Faculdade de Medicina do ABC; Mauro Bafutto, M.D, Principal Investigator — Instituto Goiano de Gastroenterologia; Carlos Fernando Francesconi, M.D, Principal Investigator — Hospital Mãe de Deus; Maria do Carmo Passos, M.D, Principal Investigator — Instituto Alfa de Gastroenterologia de BH; Flavio Steinwurtz, MD, Principal Investigator — Hospital Israelita Albert Eisntein
Locations (8):
- Brazil (8):
  - Instituto Goiano de Gastroenterologia, Goiânia, Goiás
  - Instituto Alfa de Gastroenterologia, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora das Graças, Curitiba, Paraná
  - Hospital São Lucas, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Hospital São Paulo / UNIFESP, São Paulo, São Paulo

REFERENCES:
- [Derived] Francesconi CF, Machado MB, Steinwurz F, Nones RB, Quilici FA, Catapani WR, Miszputen SJ, Bafutto M. ORAL ADMINISTRATION OF EXOGENOUS LACTASE IN TABLETS FOR PATIENTS DIAGNOSED WITH LACTOSE INTOLERANCE DUE TO PRIMARY HYPOLACTASIA. Arq Gastroenterol. 2016 Oct-Dec;53(4):228-234. doi: 10.1590/S0004-28032016000400004. PMID 27706451